CLINICAL TRIAL: NCT00266396
Title: A Randomized Trial of Weight-bearing Recommendations After Total Hip or Total Knee Arthroplasty
Brief Title: Weight-bearing Recommendation After Replacement of the Hip or Knee Joint
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Verein zur Förderung der Rehabilitationsforschung in Schleswig-Holstein (Other)
Collaborators: Verein zur Förderung der Erforschung und Bekämpfung rheumatischer Erkrankungen Bad Bramstedt e.V (Other); Landesversicherungsanstalt Schleswig-Holstein (Unknown); Landesversicherungsanstalt Freie und Hansestadt Hamburg (Unknown); Deutsche Arthrose-Hilfe (Other)
Responsible Party: Principal Investigator, Thoralf R Liebs, Consultant Orthopaedic Surgeon, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: vffr-35
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Osteoarthritis
Keywords: Total Hip Arthroplasty; THA; Total Knee Arthroplasty; TKA; Total Hip Replacement; THR; Total Knee Replacement; TKR
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- weight-bearing recommendation (Experimental): Weight-bearing recommendation after THA and TKA
  Interventions: Behavioral: Recommend full weight-bearing; Behavioral: Recommend parital weight-bearing

INTERVENTIONS:
Behavioral: Recommend full weight-bearing — The full weight-bearing group is trained in 4-point gait with crutches and is recommended to put as much weight as tolerated on the leg on which surgery has been performed, immediately after surgery
Behavioral: Recommend parital weight-bearing — The partial weight-bearing group is trained in 3-point gait with crutches and is instructed to limit weight-bearing of the affected leg to 20kg for a period of six-weeks. Scales are used to train these participants not to exceed 20kg

SUMMARY:
Despite the widespread use of total hip and knee arthroplasty, there is a notable lack of consensus regarding postoperative treatment, mostly because of the lack of well-designed studies testing the efficacy and effectiveness of such practices. In particular, there are no evidence-based recommendations on the amount of weight that the patient should be advised to bear on the operated leg after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is about to receive unilateral hip or knee replacement surgery on an elective basis for diagnosis of osteoarthritis or femoral head necrosis

Exclusion Criteria:

* A history of septic arthritis,
* Hip fracture,
* Intraoperative complications,
* History of implant surgery on the joint to be operated on,
* Rheumatoid arthritis,
* Amputations,
* Inability to complete the questionnaires because of cognitive or language difficulties.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 352
Dates: Start 2002-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Physical function, measured by means of the Western Ontario and McMaster universities (WOMAC) osteoarthritis index | Baseline, 3, 6, 12 and 24-months after surgery

SECONDARY OUTCOMES:
Leg specific stiffness and pain, both measured by the WOMAC. | Baseline, 3, 6, 12 and 24-months after surgery
Physical component summary of the SF-36 | Baseline, 3, 6, 12 and 24-months after surgery
Lequesne Hip resp. Knee Score | Baseline, 3, 6, 12 and 24-months after surgery
Patient satisfaction | Baseline, 3, 6, 12 and 24-months after surgery
Quality-Adjusted Life Years | Baseline, 3, 6, 12 and 24-months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Thoralf R Liebs, MD, Principal Investigator — University of Schleswig-Holstein Medical Center, Kiel Campus
Locations (4):
- Germany (4):
  - Ostseeklinik Damp, Department I of Orthopedic Surgery, Damp
  - University of Schleswig-Holstein Medical Center, Kiel Campus, Kiel
  - University of Schleswig-Holstein Medical Center, Lübeck Campus, Lübeck
  - Wedel Hospital, Department of Surgery, Wedel

IPD SHARING:
Plan to Share IPD: No